CLINICAL TRIAL: NCT07115147
Title: Blue Diode Laser Vaporization for BPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE2025.162
Record Dates: First submitted 2025-06-24; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: BPH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blue light laser Arm (Experimental): 450nm center wavelength blue diode 200W laser is employed for the surgical procedure
  Interventions: Device: Blue diode laser

INTERVENTIONS:
Device: Blue diode laser — All procedures would be performed under spinal or general anaesthesia. Blue diode laser vaporization would be performed according to the standard approach for the obstructing prostate

SUMMARY:
This is a prospective data collection of subjects using blude diode laser for the treatment of BPH.

DETAILED DESCRIPTION:
This is a prospective single-arm study evaluating the outcome of blue diode laser vaporization. The energy from a 450nm blue laser vaporization will be used for the treatment of BPH. The study period for each patient is 1 year. Recruited subjects will then be followed up at 3 months, 6 months and 12 months after operation. Blood tests, urine tests, ultrasound for prostate volume assessment, uroflowmetry and the same set of questionnaires will be performed again during follow-up for assessing the clinical progress. Any adverse event and unplanned admission will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 50 years
* Symptomatic BPH

Exclusion Criteria:

* Additional procedure is needed e.g. cystolithotripsy, orchidectomy etc2. Known Ca prostate patients
* Patients with history of TURP
* Known Urethral stricture / Bladder stone / Hypercontractile bladder
* Known neurological diseases which may affect bladder function (e.g. Parkinsonism, stroke) 6. Contraindicated to undergo TURP (e.g. not fit for GA/SA, active urinary tract infection, fail to be placed in lithotomy position, uncorrectable coagulopathy, antiplatelet or anticoagulant which cannot be stopped)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms measured by International Prostate Symptom Score (IPSS) score | Baseline, 1 month, 3 months, 6 months, 12 month
  Change in total scores in International Prostate Symptom Score (ranges from 0 to 35) questionnaires. The higher score, the more worse symptom
Change in urodynamic in uroflowmetry | Baseline, 1 month, 3 months, 6 months, 12 month
  Change in urodynamic function assessed by uroflowmetry

SECONDARY OUTCOMES:
Operation Time | Intra-operation
  Duration of the operation
Need of post operative irrigation | Peri-operative period
  Need of post operative irrigation
Catheter time | 1 month, 3 month, 6 month, 12 month
  Duration of catheter time in hour since completion of surgery
Hospital stay | Peri-operative period
  Duration of hospital stay in hour since completion of surgery
Transfusion rate | 1 month
  No of patient need transfusion
Verbal dysuria score | First day after catether removal
  It is assesed by a scale from 0-10; the higher score the more worse dysuria
Incidence of unplanned clinic okr hospital attendance | 90 days since completion of surgery
  Number of unplanned clinic or hospital attendance after surgery
Patient quality of life | Baseline, 1 month, 3 months, 6 months, 12 month
  Assessed with the EQ-5D-5L questionnaire from 0-100, the higher the score the better in quality of life
Erectile function measured by International Index of Erectile Function 5-item version (IIEF-5) score | Baseline, 1 month, 3 months, 6 months, 12 month
  Change in International Index of Erectile Function 5 questionnaire score (ranges from 0 to 25). The higher score, the more worse symptom
Ejaculatory function measured by MSHQ-EjD-SF (function and bother) score | Baseline, 1 month, 3 months, 6 months, 12 month
  Change in MSHQ-EjD-SF questionnaire score (Range from 1-15 for function and and 0-5 for bother). The higher score, the more worse symptom
Prostate Specific Antigen (PSA) change | Baseline, 1 month, 3 months, 6 months, 12 month
  PSA change after treatment
Adverse events (AE) and serious adverse events (SAE) related to the treatment | Baseline, 1 month, 3 months, 6 months, 12 month
  The severity of AE is grade by Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Fung Peter CHIU, MBChB PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Yee CH, Li JK, Lam HC, Chan ES, Hou SS, Ng CF. The prevalence of lower urinary tract symptoms in a Chinese population, and the correlation with uroflowmetry and disease perception. Int Urol Nephrol. 2014 Apr;46(4):703-10. doi: 10.1007/s11255-013-0586-9. Epub 2013 Oct 18. PMID 24136186
- [Background] Teoh JY, Kan CF, Tsui B, Chiu PK, Man CY, Hou SS, Ng CF. Ambulatory care program for patients presenting with acute urinary retention secondary to benign prostatic hyperplasia. Int Urol Nephrol. 2012 Dec;44(6):1593-9. doi: 10.1007/s11255-012-0266-1. Epub 2012 Aug 23. PMID 22914880
- [Background] Wei JT, Calhoun E, Jacobsen SJ. Urologic diseases in america project: benign prostatic hyperplasia. J Urol. 2008 May;179(5 Suppl):S75-80. doi: 10.1016/j.juro.2008.03.141. PMID 18405761
- [Background] Teng J, Zhang D, Li Y, Yin L, Wang K, Cui X, Xu D. Photoselective vaporization with the green light laser vs transurethral resection of the prostate for treating benign prostate hyperplasia: a systematic review and meta-analysis. BJU Int. 2013 Feb;111(2):312-23. doi: 10.1111/j.1464-410X.2012.11395.x. Epub 2012 Nov 13. PMID 23145474